CLINICAL TRIAL: NCT00643591
Title: Pilot Study on the Determination of Therapy Resistant Areas Within the Tumor in Patients With High-grade Glioma by Repeated 18F-FDG-PET-CT Scans
Brief Title: Positron Emission Tomography-Computed Tomography (PET-CT) High-grade Glioma
Status: Terminated | Type: Observational
Why Stopped: Patient compliance was low.
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MAASTRO 07-12-12/09; EudraCT Number 2007-005530-36
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Cerebral Astrocytoma, High Grade
Keywords: high grade glioma; FDG-PET-CT; blood proteins; prognosis
MeSH Terms: conditions — Astrocytoma; Glioma | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational: Patients with a primary glioblastoma
  Interventions: Other: imaging (dynamic PET-CT scan)

INTERVENTIONS:
Other: imaging (dynamic PET-CT scan) — dynamic PET-CT scan

SUMMARY:
The objectives of the trial are:

* To determine the localisation within the primary tumor of the therapy resistant cells, before and during radiotherapy to determine a possible accurate boost volume.
* To determine changes during treatment intra- and extratumoral within the irradiated area.(Intratumoral: change of up-take - decrease, increase, change of localization/ Extratumoral: effects of temporal changes in up-take - e.g. due to oedema).

DETAILED DESCRIPTION:
Patients harboring a primary intracerebral high grade tumor (WHO III- IV) have a median survival of six to 12 months. Combined chemoradiotherapy with temozolomide is now the standard of care since results of the joint EORTC-NCIC phase III study randomizing between radiotherapy alone and combined radiochemotherapy with temozolomide showed a significant improvement in 2-years survival from 8% to 24% for the combined treatment arm (Stupp 2005).

A differentiation between possible responders and non-responders before the start of irradiation may eventual be possible by the use of 18F-FDG PET-CT. Preliminary own results have shown that a higher metabolic activity in glioblastoma as measured on a simulation 18F-FDG PET-CT scan can be a prognosticator for shortened survival (Baumert, 2006).

Our preliminary data show that a high uptake of 18F-FDG on a PET-CT scan before radiotherapy in glioblastoma could be a marker for reduced survival.

Popperl et al showed that dual phase FDG PET imaging is superior in differentiating low-grade from high-grade recurrent astrocytomas (Popperl, 2006). Visual analysis of delineation of glioma showed that the delayed images (imaged first 0-90 min and once or twice later at 180-480 min after injection) better distinguished the high uptake in tumors relative to uptake in gray matter. SUV comparisons also showed greater uptake in the tumors than in gray matter, brain, or white matter at the delayed times (Spence et al).

These findings support the view that by using FDG-PET scans we could image active areas within the tumor. Indeed, in vivo, a cancer is made up by different types of cells, including hypoxic cells, cells that proliferate more fast, as well as by non-malignant tissues, including inflammatory cells and vasculature.

Intra-tumor heterogeneity in malignant glioma is often observed and can be visualised also by current PET-CT techniques.

The dynamics of the tracer uptake in the different tumor sub-volumes may give important information about the biological characteristics as well. Indeed, the dynamics of FDG uptake per cell are dependent on the blood flow, the uptake in the cell and the phosphorylation. All these of these steps give information on the biology of the cancer in that particular area of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gliomas III - IV (glioblastoma, anaplastic astrocytoma, gliosarcoma) at primary diagnosis;
* WhO PFS <= 2
* Tumours which do enhance on pre-operative imaging.
* Post-operative enough visible residual tumour on PET or status after biopsy only
* Age >18 years
* Availability of deep fresh frozen tissue for molecular biologic evaluation - if possible
* Patient able to tolerate full course of conventional RT and follow serial scanning
* No previous radiotherapy to the head and neck and brain area.
* Prior neurosurgery within 6 weeks of treatment
* No previous chemotherapy before treatment of the glioma. Standard radiochemotherapy with temozolomide is not excluded
* No prior or concurrent medical condition which would make treatment difficult to complete. Medication with steroids is allowed.
* No incapacitated patients.

Exclusion Criteria:

* Not histologically confirmed gliomas III - IV (glioblastoma, anaplastic astrocytoma, gliosarcoma) at primary diagnosis;
* WhO PFS > 2
* No tumours which do enhance on pre-operative imaging.
* Post-operative not enough visible residual tumor on PET or status after biopsy only
* Age <18 years
* No availability of deep fresh frozen tissue for molecular biologic evaluation
* Patient not able to tolerate full course of conventional RT and follow serial scanning
* Previous radiotherapy to the head and neck and brain area.
* Prior neurosurgery not within 6 weeks of treatment
* Previous chemotherapy before treatment of the glioma.
* Prior or concurrent medical condition which would make treatment difficult to complete.
* Incapacitated patients.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with radical radiotherapy for a high grade glioma.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the localisation within the primary tumour of the therapy resistant cells, before and during radiotherapy to determine the accurate boost volume. To determine changes during treatment intra- and extratumoral within the irradiated area. | after acquisition of all planned PET CTs

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta Baumert, MD PhD, Principal Investigator — Maastricht Radiation Oncology
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Netherlands